CLINICAL TRIAL: NCT03680404
Title: The Effect of Local Antioxidant Therapy on Racial Differences in Vasoconstriction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Associate Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-0441
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Vasoconstriction
Keywords: Racial Differences; Oxidative Stress
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Phenylephrine; acetovanillone; Allopurinol; tempol

STUDY DESIGN:
Intervention Model Description: Each subject has one control site and three experimental sites concurrently tested within the same study using intradermal microdialysis on the dorsal forearm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control (Phenylephrine) (Active Comparator): Subjects will be administered phenylephrine at varying concentrations (10^-2 to 10^-8 M phenylephrine) at a rate of 2 microliters/minute for 10 minutes at each dose to construct a dose-response curve.
  Interventions: Drug: Control (Phenylephrine)
- Phenylephrine + Apocynin (Experimental): Subjects will be coinfused with the same phenylephrine concentrations as the control arm and apocynin (10^-4 M) at the same rate and for the same time as the control arm.
  Interventions: Drug: Phenylephrine + Apocynin
- Phenylephrine + Allopurinol (Experimental): Subjects will be coinfused with the same phenylephrine concentrations as the control arm and allopurinol (10^-5 M) at the same rate and for the same time as the control arm.
  Interventions: Drug: Phenylephrine + Allopurinol
- Phenylephrine + Tempol (Experimental): Subjects will be coinfused with the same phenylephrine concentrations as the control arm and Tempol (10^-5 M) at the same rate and for the same time as the control arm.
  Interventions: Drug: Phenylephrine + Tempol

INTERVENTIONS:
Drug: Control (Phenylephrine) — This intervention is aimed at assessing the vascular responsiveness to phenylephrine, an alpha 1-agonist, in white and black men and women across a series of ascending dose concentrations.
  Arms: Control (Phenylephrine)
Drug: Phenylephrine + Apocynin — This intervention is meant to assess the impact of NADPH oxidase-derived superoxide on vasoconstrictor responses by inhibiting the enzyme NADPH oxidase.
  Arms: Phenylephrine + Apocynin
Drug: Phenylephrine + Allopurinol — This intervention is meant to assess the impact of xanthine oxidase-derived superoxide on vasoconstrictor responses by inhibiting the enzyme xanthine oxidase.
  Arms: Phenylephrine + Allopurinol
Drug: Phenylephrine + Tempol — This intervention is meant to assess the impact of superoxide on vasoconstrictor responses by scavenging available superoxide.
  Arms: Phenylephrine + Tempol

SUMMARY:
The goal of this study is to examine possible mechanisms of heightened vasoconstriction in Black/African American men and women as possible links to the elevated prevalence of cardiovascular dysfunction and disease. The main targets in this study are sources of oxidative stress.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) afflicts nearly one-third of the adult population with all races and ethnicities represented in CVD prevalence. Unfortunately, a disparity exists such that the black population (BL) is disproportionately affected compared to other groups, including the white population (WH). While the underlying cause of this disparity is multifactorial, vascular dysfunction (i.e., impaired vasodilation and/or augmented vasoconstriction) is a key contributor. As has been previously observed, BL exhibit a heightened vasoconstrictor response to both pharmacological (e.g., alpha-adrenergic receptor agonists) and environmental (e.g., cold pressor test) stimuli compared to their WH counterparts. Additionally, reactive oxygen species (ROS) and the subsequent reduction in nitric oxide (NO) bioavailability may partially mediate this response.

Interestingly, the small blood vessels in the skin (cutaneous microvasculature) in BL, but otherwise healthy individuals, produce an impaired blood flow response to local heating when compared to age-, body mass index (BMI)-, and gender-matched WH. However, pre-treatment of the cutaneous microvasculature with either allopurinol or apocynin (xanthine oxidase inhibitor and NADPH oxidase inhibitor, respectively) abolishes this skin blood flow difference. These drugs inhibit possible sources of ROS, which, as mentioned, may be mediating the heightened vasoconstrictor response in BL. Accordingly, apocynin administration in previous research using an animal model ameliorates alpha-adrenergic receptor-mediated vasoconstriction, possibly due to a reduction in ROS. The role of xanthine/NADPH oxidase and the production of ROS on alpha-adrenergic receptor-mediated vasoconstriction in humans remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (ages 18-35, both genders) will be recruited from the greater Arlington area to participate in the study.
* Must self-report both parents as either African American or Caucasian American.

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, than we may still opt to proceed with data collection.
* Individuals with cardiovascular, neurological, and/or metabolic illnesses will be excluded from participating as well as individuals with a history of various diseases of the microvasculature including Reynaud's disease, cold-induced urticaria, cryoglobulinemia, etc.
* Subjects currently taking any prescription medications and individuals with a body mass index about 30 kg/m2) will be excluded.
* Pregnant subjects and children (i.e. younger than 18) will not be recruited for the study. Eligible females will be scheduled for days 2-7 of their menstrual cycle to account for hormonal effects on blood flow. A regular menstrual cycle is required to identify and schedule the study for the low hormone period, therefore females who lack a regular cycle will be excluded from the study. Females currently taking birth control are eligible, as long as they can be scheduled during a low-hormone "placebo" week. If their hormone do not contain a placebo week than these individuals will not be eligible for data collection. Females who are breast-feeding will also be eligible as there are no systemic or lasting effects of the proposed vasoactive agents.
* Given that smoking can affect the peripheral vasculature, current smokers and individuals who regularly smoked (>1 pack per two weeks) within the prior 2 years will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Vasoconstrictor Responsiveness to Phenylephrine using Laser Doppler Fluxmetry | Through study completion, an average of 1 Year
  Establish heightened vasoconstriction to phenylephrine stimulation in black men and women with a focus on black women. Following local infusions of phenylephrine, the changes in blood flux will be quantified using laser Doppler fluxmetry. All changes in flux will be normalized and reported as a percentage of baseline flux.
Role of Oxidative Stress in Heightened Vasoconstriction using Laser Doppler Fluxmetry | Through study completion, an average of 1 Year
  Determine to what degree superoxide, either generally available or produced through xanthine/NADPH oxidases, contributes to heightened phenylephrine-mediated vasoconstriction. Following local coninfusions of phenylephrine with apocynin, allopurinol, or tempol, the changes in blood flux will be quantified using laser Doppler fluxmetry. All changes in flux will be normalized and reported as a percentage of baseline flux.

CONTACTS AND LOCATIONS:
Locations (1):
- Science and Engineering Research and Innovation Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No